CLINICAL TRIAL: NCT00178932
Title: Improving Outcome in Schizophrenia Through Identification of Genetic Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9132
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depression
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Outcome in schizophrenia with certain antipsychotic (Active Comparator): clozapine
  Interventions: Procedure: genetic analysis; Procedure: genetic assay
- 2 Outcome in schizophrenia with other Antipsychotics (Active Comparator): Other Antipsychotics
  Interventions: Procedure: genetic analysis; Procedure: genetic assay

INTERVENTIONS:
Procedure: genetic analysis — genetic assay of blood sample drawn with patient's consent
Procedure: genetic assay — genetic assay of blood sample drawn with patient's consent

SUMMARY:
The goals of this study are to replicate previous findings of genetic predictors of response to clozapine and other antipsychotic drugs.

ELIGIBILITY:
Inclusion Criteria:

Patients with the diagnoses of schizophrenia or schizoaffective disorder, and bipolar disorder or major depression with psychotic features, or volunteers with no history of a psychotic disorder.

Exclusion Criteria:

Patients with DSM-IV diagnoses other than schizophrenia or schizoaffective disorder, and bipolar disorder or major depression with psychotic features.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1998-11 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
We plan to compare the polymorphisms across schizophrenic patients and adults who do not have a diagnosed major mental illness. . | single visit

SECONDARY OUTCOMES:
We will also evaluate relationships between the polymorphism and past and current mental health among the non-diagnosed sample | single visit

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Y Meltzer, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Psychiatric Hospital at Vanderbilt, Nashville, Tennessee, United States